CLINICAL TRIAL: NCT01543724
Title: A Multimodal Brain Imaging Study to Investigate Neural Correlates for Therapeutic Mechanisms of Lithium in Bipolar Disorder: Glycogen Synthase Kinase 3β Single Nucleotide Polymorphisms and Gray Matter Volume Increase Following Lithium Treatment in Bipolar Disorder
Brief Title: Neural Correlates for Therapeutic Mechanisms of Lithium in Bipolar Disorder
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: The research project has been cancelled before any participants were enrolled.
Sponsor: Ewha Womans University (Other)
Collaborators: Soon Chun Hyang University (Other)
Responsible Party: Principal Investigator, In Kyoon Lyoo, Professor, Ewha Womans University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: bpli2008
Record Dates: First submitted 2012-02-28; First posted 2012-03-05 (Estimated); Last update posted 2018-02-09 (Actual); Status verified 2018-02

CONDITIONS: Bipolar Disorder
Keywords: Lithium; Bipolar disorder; Multimodal Brain Imaging
MeSH Terms: conditions — Bipolar Disorder | interventions — Lithium

ARMS (1):
- Lithium (Experimental)
  Interventions: Drug: Lithium

INTERVENTIONS:
Drug: Lithium — 10mg/kg/day for 12 weeks

SUMMARY:
The investigators will assess Li-induced gray matter volume changes with regard to the endophenotype of GSK3beta polymorphism. The changes of gray matter are supposed to be more attributable to neurotrophic and neuroprotective characteristics of Li, which were closely related to the inhibition of apoptotic activity of GSK3beta.

ELIGIBILITY:
Inclusion Criteria:

* Men and Women aged between 19 and 55
* Diagnosis of bipolar I disorder as assessed by the structured clinical interview for DSM-IV (SCID-IV)
* Patients who have not used psychoactive medications for more than 2 weeks
* Individuals who provided written consent for participation

Exclusion Criteria:

* Presence of any major physical or neurological illness (e.g., head trauma, epilepsy, seizure, stroke, cerebral tumor, multiple sclerosis, cerebrovascular disease, narrow-angle glaucoma, drug hypersensitivity, etc.)
* Women who are pregnant, breastfeeding, or planning pregnancy
* Diagnosis of any Axis I disorder other than bipolar disorder
* Intelligence quotient below 80
* Current or past drug abuse
* Contraindications to magnetic resonance imaging (e.g., pacemaker implantation, claustrophobia, etc.)

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2015-06-01 (Estimated); Primary Completion 2017-12-31 (Estimated); Study Completion 2017-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in manic symptom scores at 12 weeks | Baseline and at 12 weeks
Change from baseline in manic symptom scores at 8 weeks | Baseline and at 8 weeks
Change from baseline in manic symptom scores at 4 weeks | Baseline and at 4 weeks
Change from baseline in manic symptom scores at 1 week | Baseline and at 1 week
Change from baseline in depressive symptom scores at 12 weeks | Baseline and at 12 weeks
Change from baseline in depressive symptom scores at 8 weeks | Baseline and at 8 weeks
Change from baseline in depressive symptom scores at 4 weeks | Baseline and at 4 weeks
Change from baseline in depressive symptom scores at 1 week | Baseline and at 1 week
Change from baseline in global function scores at 12 weeks | Baseline and at 12 weeks
Change from baseline in global function scores at 8 weeks | Baseline and at 8 weeks
Change from baseline in global function scores at 4 weeks | Baseline and at 4 weeks
Change from baseline in global function scores at 1 week | Baseline and at 1 week

SECONDARY OUTCOMES:
Changes from baseline in brain structure analyzed using computational approach | Baseline and at 12 weeks
Number of participants with adverse events | 12 weeks
Number of participants with adverse events | 8 weeks
Number of participants with adverse events | 4 weeks
Number of participants with adverse events | 1 week

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea